CLINICAL TRIAL: NCT02037373
Title: Post-Marketing Requirement Study to Evaluate the Safety of Octaplas™ Versus Plasma in Patients Undergoing Orthotopic Liver Transplantation With Special Emphasis on Hyperfibrinolysis.
Brief Title: Evaluation of the Safety of Octaplas™ Versus Plasma in Patients Undergoing Orthotopic Liver Transplantation
Status: Terminated | Type: Observational
Why Stopped: FDA released requirement to complete study
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: LAS-215
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Coagulopathy; Endstage Liver Disease
Keywords: intra and post-op coagulopathy in patients undergoing OLT
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Octaplas™: Patients treated with Octaplas™ infusion solution for IV administration as prescribed by their treating physician.
  Interventions: Biological: Octaplas™
- Plasma: Patients treated with regular plasma (e.g., fresh frozen plasma (FFP) and other FDA and American Association of Blood Banks (AABB) approved plasma products).
  Interventions: Biological: Plasma

INTERVENTIONS:
Biological: Octaplas™ — Octaplas™ infusion solution for IV administration as prescribed by the treating physician.
  Groups: Octaplas™
Biological: Plasma — Plasma as prescribed by the treating physician.
  Other Names: FFP and other approved plasma products
  Groups: Plasma

SUMMARY:
Post-Marketing Requirement study to evaluate the safety of octaplas™ versus plasma in patients undergoing orthotopic liver transplantation (OLT). The primary objective is to assess the incidence of hyperfibrinolysis in patients undergoing (OLT) receiving octaplas™ versus regular plasma (e.g., fresh frozen plasma and other FDA and AABB approved plasma products).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥18 years
* Patient is scheduled to undego orthotopic liver transplantation (OLT)
* Patient has a natural MAYO End-Stage Liver Disease (MELD) score of 15-40
* Patient is willing to give voluntary written informed consent before any study- related procedure is to be performed that is not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudicing future medical care

Exclusion Criteria:

* Patient has a history of severe hypersensitivity reaction to plasma-derived products or to any excipient of the investigational product
* Patient is known to be IgA deficient with documented antibodies against IgA
* Patient is a planned recipient for a living donor OLT
* Patient has a severe deficiency of Protein S
* Patient is currently participating in an interventional clinical study or has participated in one within 30 days of the date of their OLT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include patients undergoing orthotopic liver transplantation
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-08; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
To assess the incidence of hyperfibinolysis in patients undergoing OLT receiving octaplas™ versus regular plasma (e.g., fresh frozen plasma (FFP) and other FDA and American Association of Blood Banks (AABB) approved plasma products). | 3 days (perioperative period plus post-operative follow-up)
  The incidence of 'clinically relevant hyperfibrinolytic events' in patients receiving octaplas™ will be compared with the incidence rate in patients receiving plasma. For this trial a 'clinically relevant hyperfibrinolytic event' is defined as a decrease of at least 7.5% in the maximum amplitude (MA) as measured by the thromboelastography (TEG) or rotational thromboelastography (ROTEM) within 30 minutes after MA is achieved and the event is associated with bleeding requiring intervention.

SECONDARY OUTCOMES:
The safety of octaplas™ in comparison to plasma will be assessed by monitoring the occurrence of adverse drug reactions (i.e., transfusion reactions). | 3 days (perioperative period plus post-operative follow-up)
  The incidence of all adverse drug reactions (i.e., transfusion reactions) during the study period among patients receiving octaplas™ in comparison to standard plasma products.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, Study Director — International Medical Monitor
Locations (4):
- United States (4):
  - Octapharma Research Site, Loma Linda, California
  - Octapharma Research Site, Philadelphia, Pennsylvania
  - Octapharma Research Site, Pittsburgh, Pennsylvania
  - Octapharma Research Site, Nashville, Tennessee